CLINICAL TRIAL: NCT06481358
Title: Study Using Deep Learning-based Artificial Intelligence for the Diagnosis of Small Bowel Obstruction
Brief Title: Deep Learning-based Artificial Intelligence for the Diagnosis of Small Bowel Obstruction
Status: Active, not recruiting | Type: Observational
Sponsor: Nagoya University (Other)
Responsible Party: Principal Investigator, Aitaro Takimoto, Medical Staff, Nagoya University
Other Study IDs: 2022-0188
Record Dates: First submitted 2024-06-25; First posted 2024-07-01 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Bowel Obstruction; Artificial Intelligence
MeSH Terms: conditions — Intestinal Obstruction | interventions — Artificial Intelligence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AI group: Participants read CT images with AI.
  Interventions: Diagnostic Test: Artificial intelligence
- Manual group: Participants read CT images without AI

INTERVENTIONS:
Diagnostic Test: Artificial intelligence — AI extract intestinal region and reconstruct into 3D image.
  Groups: AI group

SUMMARY:
The study will compare the diagnostic accuracy and time to diagnosis of computed tomography images of patients with suspected intestinal obstruction seen in the emergency room by residents and surgeons, with and without artificial intelligence.

DETAILED DESCRIPTION:
DESIGN: This is an diagnostic study. SETTING: We developed a deep learning-based AI technology to automatically extract the intestinal tract from CT images using 5 200 CT images of 158 patients. The CT images of patients who visited the emergency department and were suspected of small bowel obstruction between June 6 and July 26, 2018, were obtained from two tertiary referral centers, which were used as the test samples. Data analysis was completed in December 2023.

PARTICIPANTS: Residents and surgeons participated in the study. INTERVENTIONS: Residents and surgeons were divided into two groups: one group read using the AI technology, and the other group read without the AI technology.

MAIN OUTCOMES AND MEASURES: Participants indicated whether or not small bowel obstruction and obstruction location. The time for diagnosis was also collected. We applied a hierarchical Bayesian model.

ELIGIBILITY:
Inclusion Criteria:

* Persons with documented consent

Exclusion Criteria:

* Persons without documented consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 20 people
Sampling Method: Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-06-06 (Actual); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
The diagnosis of the obstruction site | September, 2024
  Accuracy of diagnosis of the obstruction site

CONTACTS AND LOCATIONS:
Overall Officials: Hieoo Uchida, PhD., Study Chair — Nagoya University Graduate School of Medicine, Pediatric Surgery
Locations (1):
- Nagoya University Graduate School of Medicine, Nagoya, Aichi-ken, Japan

IPD SHARING:
Plan to Share IPD: No